# **Informed consent form for adult above 21 years of age, for the study:**

A Comparative Study of Two Dry Needling Interventions for Plantar Heel Pain

Clinical trial: NCT03236779

Author: ZAID ALBOLOUSHI

DATE: 23-01-2021

#### Informed Consent Form for adult above 21 years of age

### أقرار مستنير (للبالغين كاملى الاهلية 21 سنة فأكثر)

إسم الباحث د زيد حبيب البلوشي

عنوان البحث: Managements Of Plantar Fasciitis Using Self-Stretching And Dry Needling عنوان البحث: Therapy

APhysical Medicine and Rehabilitations (Physical Therapy Department) مكان إجراء البحث: Hospital Kuwait

أنت مدعو(ة) للمشاركة ببحث علمي سريري سيجرى في مستشفى الطب الطبيعي و التأهيل الصحي. الرجاء أن تأخذ(ي) الوقت الكافي لقراءة المعلومات التالية بتأن قبل أن تقرر(ي) إذا كنت تريد(ين) المشاركة أم لا. بإمكانك طلب إيضاحات أو معلومات إضافية عن أي شيء مذكور في هذه الإستمارة أو عن هذه الدراسة.

تقييم طريقة العلاج الطبيعي للمرضى الذين يعانون من التهاب في أغشية باطن القدم و ذلك بهدف تطوير البروتوكولات العلاجية:

- 1- لك كامل الحرية في المشاركة أو عدم المشاركة في هذا البحث لان المشاركة ( أختيارية ).
- 2- في حالة عدم المشاركة يمكنك الانسحاب من الدراسة (البحث) في اي وقت دون أبداء الاسباب في حالة عدم المشاركة أو الانسحاب من الدراسة. و ذلك لايؤثر في حقك الكامل للرعاية الصحية المقررة لك.
- 3- في حالة الموافقة يتعهد الباحثون بالمحافظة على خصوصية و سرية المعلومات و لن يتم تداولها خارج نطاق البحث و سيتم التعامل مع النتائج لغرض البحث فقط.
- 4- في حالة المشاركة في البحث فأن أختصاصي الباحث سيقوم بأجراء مقابلة شخصية معك لتقييم حالتك الصحية و تعباءة النموذج الخاص بالدراسة مع مراعاة الخصوصية الكاملة.

لا يسمح بالمشاركة في هذة الدراسة:

- ✓ النساء الحوامل
- المرضى تحت سن القانوني او فوق سن ال 60 سنة
- ◄ المرضى الذين يعانون من مشاكل قلبية (عدم انتضام ضربات القلب، بطارية في القلب،)
  - ﴿ المرضى الذين يعانون من كسور في نفس جهة الاصابة
    - ﴿ المرضى الذين يعانون من أمراض الروماتيزم
      - ﴿ المرضى الذين يعانون من هشاشة العظام
  - ◄ المرضى الذين تم عمل عملية لا ألتهاب أغشية باطن القدم منذ 6 أشهر.



### أ. وصف البحث العلمي وهدفه وتفسير مجرياته

الوخز بالابر الجاف

. الوخز بالابر الجافة يعتبر من العلاجات الحديثة نسبيا و هي تختلف عن العلاج بالطب الصيني ولكن تحمل نفس الخاصية من حيث ان الابر لا تحمل اي محلول دوائي،الابر الجافة تستخدم أبر خيطية خالية من اي دواء او مشتقاته (مشابهة للابر الصينية) و تستخدم للعضلات الليفية التي تشكل في العضلات و تسبب العقد العضلية في التعبير العام (قولوني) و بهذه الطريقة يتم تحفيز العضلة و أزالة الشد العضلي .

الشكوى الأكثر شيوعا بعد جلسة الوخر بالابر وعادة ما يكون ووجع العضلات كمثال بعض تمرين رياضي شديد. هذه المشاعر عادة ما تهدأ بعد بعد 24 أو 48 ساعة ، جنبا إلى جنب مع الألم الأصلي قبل العلاج الوخر بالابر

- 1- بعض الالم بعد الجلسة.
- 2- الحساسية من الابر للبعض المرضى
- 3- الكدمات التي قد تصاحب في بعض الاحيان و بعض المناطق
- 4- احتمالية بسيطة لحصول الأسترواح الرئوي (بعض عضلات الصدر القريبة من الرئة).
  - 5- احتمالية حالة الهبوط في ضغط الدم او الغثيان.

### ب. اذكر الفوائد التي قد تنتج عن هذا البحث:

الوخز بالابر الجافة هو إجراء فريد من نوعه يهدف خصيصا لاستهداف واستعادة وظيفة العضلات، مع التركيز على تحسين شفاء الأنسجة واستعادة وظيفة الأنسجة الطبيعية. هذا أمر مهم لاستمرار النشاط مع وظيفة العضلات الفقيرة قد يؤدي إلى مزيد من تلف الأنسجة وزيادة الألم. وليس المقصود الوخز بالابر الجافة لتحل محل الإجراءات الطبية التقليدية مثل العلاج الطبيعي أو الجراحة. ومع ذلك، فانها طريقة تعمل جنبا إلى جنب مع خيارات العلاج التقليدي، يمكن أن الوخز بالابر الجافة تكون وسيلة مؤثرة لتسريع الحد من الألم، وتضميد الجراح واستعادة وظيفة الأنسجة الطبيعية.

في حال وافقت على المشاركة في هذه الدراسة، سيبقى إسمك طي الكتمان. لن يكون لأي شخص، ما لم ينص القانون على ذلك، حق الإطلاع على ملفك الطبي باستثناء الباحثون و الطبيب المسوؤل عن حالتك الصحية و المسؤلون عن الدراسة ومعاونيه، ولجان الأخلاق المهنية المستقلة، و مفتشين من اللإدارات الحكومية المنظمة.



### في حالة الموافقة سيتم أستخدام أسلوب:

- 1- الابر الجافة المعقمة
- 2- المكان الذي سيتم علاجه هو عضلات القدم و الساق
- 3- العلاج سيتكون من 8 جلسات بمعدل جلسة او جلستين في الاسبوع مدة العلاج ستكون شهر.
- 4- لا يتضمن هذا البحث أعطائ اي أدوية أو اجراء تجارب طبية أو اخذ عينة حيوية من المريض أو تعديل البوتوكولات العلاجية.

#### موافقة المشترك:

لقد قرأت استمارة القبول هذه وفهمت مضمونها. تمت الأجابة على أسئلتي جميعها. وبناء عليه فأنني، حرا مختارا، أجيز إجراء هذا البحث و أوافق على الإشتراك فيه، وإني أعلم ان الباحث الدكتور زيد حبيب البلوشي. وزملاءه ومعاونيه او مساعديه سيكونون مستعدين للإجابة على أسئلتي، وأنه باستطاعتي الإتصال بهم على الهاتف 55079760. وإذا شعرت لاحقا ان الأجوبة تحتاج الى مزيد من الإيضاح فسوف أتصل بأحد اعضاء لجنة الأخلاقيات.

كما أعرف تمام المعرفة بانني حرفي الإنسحاب من هذا البحث متى شئت حتى بعد التوقيع على الموافقة دون ان يؤثر ذلك على العناية الطبية المقدمة لي. أعلم أني سوف أحصل على نسخة طبق الأصل عن هذه الموافقة.

الاسم:

٥ موافق:

التوقيع:

التاريخ:

و لا أوافق:



الاسم:

التوقيع:

التاريخ:

## Dar Almaajim International Translation **Typing Photocopying Company**



# وطباعة وتصوير المستندات

## Informed Consent Form for adult above 21 years of age

Researcher's name: Dr. ZAID HABIB AL-BOLOUSHI

Research title: Managements of Plantar Fasciitis Using Self-Stretching and Dry

Needling Therapy

Place of research: (Physical Therapy Department) Physical Medicine and

Rehabilitations Hospital Kuwait

You are invited to participate in clinical scientific research that will be conducted at the Physical Medicine and Health Rehabilitation Hospital. Please take the time to carefully read the following information before deciding whether or not you want to participate. You can request additional clarifications or information about anything mentioned in this form or about this study.

Evaluating the physiotherapy method for patients suffering from inflammation of the sole of the foot membranes with the aim of developing treatment protocols:

1- You are completely free to participate or not participate in this research

because participation is (optional).

2- In case of non-participation, you can withdraw from the study (research) at any time without giving reasons in case of non-participation or withdrawal from the study. This does not affect your full right to the health care prescribed to you.

3- In case of approval, the researchers shall undertake to maintain the privacy and confidentiality of the information, and it will not be circulated outside the scope of the research, and the results will be treated for the purpose of the

research only.

4- In case that of your participation in the research, the researcher's specialist will conduct a personal interview with you to assess your health condition and fill out the study form, taking into account complete privacy.

It is not allowed to the following to participate in the study:

> Pregnant women

> Patients under the legal age or over the age of 60 years

> Patients with cardio problems (arrhythmias, battery in the heart)

> Patients with fractures on the same side of the injury

> Patients with rheumatic diseases

> Patients with osteoporosis

> Patients who underwent an operation for sole of the foot membranes inflammation since 6 months.

Mg.



## Dar Almaajim International Translation Typing Photocopying Company



### شركه دار المعاجم الدولية للترجمة وطباعة وتصوير المستندات

A- Description of scientific research and its goal and interpretation of its course Dry needling

Dry needling is considered a relatively modern treatment and it differs from Chinese medicine treatment, but it has the same feature, that the needles do not carry any medicinal solution, dry needles use threaded needles free of any medicine or its derivatives (similar to Chinese needles) and are used for muscle fibers that It forms in the muscles and causes the muscle nodes in the general expression (colonic), and in this way the muscle is stimulated and the muscle strain is removed.

The most common complaint after needling session is usually muscle soreness, for example, some vigorous exercise. These feelings usually subside after 24 or 48 hours, along with the original pain before needling treatment.

- 1- Some pain after the session.
- 2- Allergy from needles for some patients
- 3- Bruises that may accompany in some cases and in some areas
- 4- A slight chance of pneumothorax (some chest muscles close to the lung).
- 5- The possibility of a state of low blood pressure or nausea.

### B- Mention the benefits that may result from this research:

Dry needling is a unique procedure specifically designed to target and restore muscle function, with an emphasis on improving tissue healing and restoring normal tissue function. This is important for activity continuity with poor muscle function may lead to further tissue damage and increased pain. Dry needling is not intended to replace traditional medical procedures such as physical therapy or surgery. However, it is a method that works in conjunction with traditional treatment options, dry needling can be an effective way to accelerate pain reduction, heal wounds and restore normal tissue function.

If you agree to participate in this study, your name will be kept confidential. No person, unless required by law, will have the right to view your medical file, except for researchers, the doctor in charge of your health, the study officers and his assistants, independent professional ethics committees, and inspectors from organized government departments.

THE THE WINDS AND PHOTOGRAPH OF THE PROPERTY O

Ma,

Dar Almaajim Intl. Translation, Typing & Photocopying Company Salmiya, Salem Al Mubarak Street, after AUK

8Mall, Mezanine Floor, Office No.13, CR 408212

شركه دار المعاجم الدولية للترجمة وطباعة وتصوير المستندات السالمية، شارع سالم المبارك، بعد الجامعة الأمريكية بالكويت، إيت مول، دور ميزانين، مكتب رقم (13). سجل تجاري (408212)

## Dar Almaajim International Translation Typing Photocopying Company



### شركه دار المعاجم الدولية للترجمة وطباعة وتصوير المستندات

In case of approval, the method will be used:

1- Sterile dry needles

2- The part to be treated is the leg and leg muscles

3- The treatment will consist of 8 sessions, an average of one or two sessions per week, and the duration of treatment will be one month.

4- This research does not include giving any drugs, conducting medical experiments, taking vital samples from patients, or modifying treatment protocols.

Acceptance of the participant:

I have read this acceptance form and understand its content. All my questions have been answered. Accordingly, I, with my own capacity, hereby authorize this research and agree to participate in it, and I know that the researcher, Dr. ZAID HABIB ALBOLOUSHI, his colleagues and his assistants or associates will be ready to answer my questions, and that I can contact them on the phone 55079760. If I feel later that the answers require further clarification, I will contact a member of the Ethics Committee.

I also know very well that I am free to withdraw from this research whenever I want even after signing the approval without affecting the medical care provided to me. I know that I will receive an exact copy of this approval.

| o Agree | Name |
|---------------|-----------|
| | Signature |
| | Date: |
| o Don't agree | Name |
| | Signature |
| | Date |

Ma.



شركه دار المعاجم الدولية للترجمة وطباعة وتصوير المستندات السامية، شارع سالم المبارك، بعد الجامعة الأمريكية بالكويت، إيت مول، دور ميزانين، مكتب رقم (13). سجل تجارى (408212)